CLINICAL TRIAL: NCT04830371
Title: A Phase II/III, Multicenter, Observer-Blinded, Randomized, Non-inferiority and Safety Study of Typhoid Conjugate Vaccine (EuTCV) Compared to Typbar-TCV in Healthy 6 Months-45 Years Aged Participants
Brief Title: Non-inferiority and Safety Study of EuTCV Compared to Typbar-TCV in Healthy 6 Months-45 Years Aged Participants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EuVCT_TCV301
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-03

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Vi-CRM197, Batch #1) (Experimental): Single dose of Typhoid Conjugate Vaccine (Vi-CRM197) Batch #1 will be intramuscularly administered at Day 0.
  Interventions: Biological: EuTCV (Vi-CRM Typhoid conjugate vaccine)
- Arm A (Vi-CRM197, Batch #2) (Experimental): Single dose of Typhoid Conjugate Vaccine (Vi-CRM197) Batch #2 will be intramuscularly administered at Day 0.
  Interventions: Biological: EuTCV (Vi-CRM Typhoid conjugate vaccine)
- Arm A (Vi-CRM197, Batch #3) (Experimental): Single dose of Typhoid Conjugate Vaccine (Vi-CRM197) Batch #3 will be intramuscularly administered at Day 0.
  Interventions: Biological: EuTCV (Vi-CRM Typhoid conjugate vaccine)
- Arm D (Typbar-TCV) (Active Comparator): Single dose of Typhoid Conjugate Vaccine (Typbar-TCV) will be intramuscularly administered at Day 0.
  Interventions: Biological: Typbar-TCV

INTERVENTIONS:
Biological: EuTCV (Vi-CRM Typhoid conjugate vaccine) — Single dose, Intramuscular administration
  Arms: Arm A (Vi-CRM197, Batch #1); Arm A (Vi-CRM197, Batch #2); Arm A (Vi-CRM197, Batch #3)
Biological: Typbar-TCV — Single dose, Intramuscular administration
  Arms: Arm D (Typbar-TCV)

SUMMARY:
This is an observer-blinded, comparative, single dose, clinical phase II/III study to assess the immunogenicity and safety of EuTCV compared to Typhoid conjugate vaccine in healthy Filipino participants aged 6 months to 45 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy participants ≥6 months and ≤45 years of age at enrolment
2. Participants/Parents/Legally Authorized Representative(LAR) willing to give written informed consent/assent to participate in the trial
3. Participants/Parents/LAR willing to follow the study procedures of the study and available for the entire duration of the study
4. Participants who are healthy as determined by medical history, with no clinically significant abnormalities in clinical examination and laboratory tests
5. Female participants must have a negative serum (at Screening) and negative urinary (at Day 1) pregnancy test and agree to use 2 methods of contraception from dosing until 90 days after vaccination.

Exclusion Criteria:

1. Participants/Parents/LAR unwilling to give his/her consent/assent to participate in the trial
2. Participants concomitantly enrolled or scheduled to be enrolled in another trial
3. Children and infants with a congenital abnormality
4. Known history of immune function disorders including immunodeficiency disease, or chronic use of systemic steroids, cytotoxic or other immunosuppressive drugs
5. Pregnant, lactating women or women of childbearing age not using a reliable method of contraception
6. History of uncontrolled coagulopathy or blood disorders
7. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the participant and interfere with the assessment of the trial objectives
8. History of alcohol or substance abuse

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 444 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 4 weeks after vaccination of EuTCV (pooled of 3 batches)/Typbar-TCV compared to baseline
Proportion of Solicited local and systemic AEs | 7 days after vaccination
Proportion of unsolicited AEs | within 28 days after vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- Philippines (2):
  - De La Salle Medical and Health Sciences Institute, Cavite
  - University of the East Ramon Magsaysay Memorial Medical Center, Quezon City

REFERENCES:
- [Derived] Ok Baik Y, Lee Y, Lee C, Kyung Kim S, Park J, Sun M, Jung D, Young Jang J, Jun Yong T, Woo Park J, Jeong S, Lim S, Hyun Han S, Keun Choi S. A Phase II/III, Multicenter, Observer-blinded, Randomized, Non-inferiority and Safety, study of typhoid conjugate vaccine (EuTCV) compared to Typbar-TCV(R) in healthy 6 Months-45 years aged participants. Vaccine. 2023 Mar 3;41(10):1753-1759. doi: 10.1016/j.vaccine.2022.12.007. Epub 2023 Feb 9. PMID 36774331